CLINICAL TRIAL: NCT00541242
Title: Safety and Efficacy of Bimatoprost Compared With Latanoprost in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-034
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-09

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Bimatoprost; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): bimatoprost 0.03% eye drops
  Interventions: Drug: bimatoprost 0.03% eye drops
- 2 (Active Comparator): latanoprost 0.005% eye drops
  Interventions: Drug: latanoprost 0.005% eye drops

INTERVENTIONS:
Drug: bimatoprost 0.03% eye drops — Open-labeled latanoprost 0.005% 1 drop into each eye every evening for 6 weeks followed by a masked randomized treatment of bimatoprost 0.03% 1 drop every evening for 12 weeks
  Other Names: latanoprost = Xalatan®; bimatoprost = Lumigan®
  Arms: 1
Drug: latanoprost 0.005% eye drops — Open-labeled latanoprost 0.005% 1 drop into each eye every evening for 6 weeks followed by a masked randomized treatment of latanoprost 0.005% 1 drop every evening for 12 weeks
  Other Names: Xalatan®
  Arms: 2

SUMMARY:
The study will compare the safety and efficacy of Bimatoprost and Latanoprost in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or chronic glaucoma
* Patient requires IOP-lowering therapy in both eyes

Exclusion Criteria:

* Uncontrolled medical conditions
* Hypersensitivity to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimatoprost 0.03% Eye Drops: Bimatoprost 0.03% eye drops
- Latanoprost 0.005% Eye Drops: Latanoprost 0.005% eye drops
Period: Treatment Period 1
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops
Started | 0 | 586 (586 patients were enrolled and received open-label latanoprost for 6 weeks)
Completed | 0 | 586 (43 of the 586 patients did not enter Treatment Period 2 (Randomized at Week 6))
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops
Started | 270 | 273
Completed | 261 | 266
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops | Total
Number analyzed (Participants) | 270 | 273 | 543
Age, Customized [Number; unit: participants] — Intent to Treat (ITT) population used for Baseline characteristics. The ITT population included all patients who were randomized (started Treatment Period 2)
  participants
    < 45 years | 9 | 16 | 25
    Between 45 and 65 years | 111 | 120 | 231
    > 65 years | 150 | 137 | 287
Sex: Female, Male [Count of Participants; unit: Participants] — Intent to Treat (ITT) population used for Baseline characteristics. The ITT population included all patients who were randomized (started Treatment Period 2)
  Participants
    Female | 147 | 155 | 302
    Male | 123 | 118 | 241

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP) at Week 12
Description: Change from Baseline in mean diurnal IOP. IOP is a measurement of the fluid pressure inside the eye. Mean diurnal IOP is the average of the IOP values of both eyes at each time point measured at 8AM, 12PM and 4PM. For each eye, the IOP was either the average of the 2 measurements, or, if a third measurement was required, the median of the 3 measurements. A negative number change from Baseline indicated a reduction in IOP.
Time Frame: Baseline, Week 12
Population: Modified Intent-to-Treat (m-ITT). The m-ITT population included all patients who started the study (randomized) and had at least a baseline and one follow-up visit measurement of IOP after receiving the study medication.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops
Number analyzed (Participants) | 270 | 272
millimeters of mercury (mmHg)
  Baseline | 21.90 (3.656) | 22.16 (3.569)
  Week 12 | -5.64 (2.968) | -4.89 (2.872)

2. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP) at Week 18
Description: as for outcome 1
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops
Number analyzed (Participants) | 270 | 272
millimeters of mercury (mmHg)
  Baseline | 21.90 (3.656) | 22.16 (3.569)
  Week 18 | -5.77 (3.023) | -5.09 (2.709)

ADVERSE EVENTS:
Description: SAEs and other AEs in the Latanoprost(LAT) Arm include those events reported by pts who received LAT in Treatment Period 1 AND those who were randomized to and received LAT in Treatment Period 2. SAEs and other AEs in the Bimatoprost(BIM) Arm only include those events reported for pts who were randomized to and received BIM in Treatment Period 2.
Arm/Group | Bimatoprost 0.03% Eye Drops | Latanoprost 0.005% Eye Drops
Serious Adverse Events (participants affected / at risk) | 4/269 | 11/586
Other Adverse Events (participants affected / at risk) | 59/269 | 89/586
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Eye Drops (N=269) | Latanoprost 0.005% Eye Drops (N=586)
Cellulitis (Infections and infestations) | 0 | 1 — Event occurred in Treatment Period 1
Coronary artery disease (Cardiac disorders) | 0 | 1 — Event occurred in Treatment Period 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 — The 2 SAEs in the Latanoprost arm occurred in Treatment Period 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Event occurred in Treatment Period 1
Aortic anyeurysm (Vascular disorders) | 0 | 1 — Event occurred in Treatment Period 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 — Event occurred in Treatment Period 1
Prostamegaly (Reproductive system and breast disorders) | 0 | 1 — Event occurred in Treatment Period 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Eye Drops (N=269) | Latanoprost 0.005% Eye Drops (N=586)
Conjunctival hyperaemia (Eye disorders) | 59 | 89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo